CLINICAL TRIAL: NCT01827553
Title: Significance of Chemoradiation Following Induction Chemotherapy in Locally Advanced,Unresectable Pancreatic Cancer -a Randomised Phase 3 Trial: Chemoradiation Following Induction Chemotherapy Compared With Chemotherapy Alone
Brief Title: Pancreatic Carcinoma: Chemoradiation Compared With Chemotherapy Alone After Induction Chemotherapy
Acronym: CONKO-007
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2009-014476-21
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Last update posted 2024-04-11 (Actual); Status verified 2023-08

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; chemoradiotherapy; chemotherapy; FOLFIRINOX; gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Induction Chemotherapy; Gemcitabine; folfirinox; Radiotherapy; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Induction CT, chemoradiotherapy (Experimental): Induction chemotherapy with gemcitabine or FOLFIRINOX; Radiotherapy, 28 x 1.8 Gy; Chemotherapy, gemcitabine;
  Interventions: Drug: Induction chemotherapy with gemcitabine or FOLFIRINOX; Radiation: Radiotherapy, 28 x 1.8 Gy; Drug: Chemotherapy, gemcitabine
- Induction CT, chemotherapy (Active Comparator): Induction chemotherapy with gemcitabine or FOLFIRINOX; Chemotherapy with gemcitabine or FOLFIRINOX according to induction chemotherapy
  Interventions: Drug: Induction chemotherapy with gemcitabine or FOLFIRINOX; Drug: Chemotherapy with gemcitabine or FOLFIRINOX according to induction chemotherapy

INTERVENTIONS:
Drug: Induction chemotherapy with gemcitabine or FOLFIRINOX — According to medical recommendation, induction chemotherapy is performed with gemcitabine (3 cycles a 3 administrations, 1000 mg/m^2/d)or FOLFIRINOX (6 cycles; 1 cycle: oxaliplatin 85 mg/m^2 2 h infusion, folinic acid 400 mg/ m^2 2h infusion completed after 30 min with irinotecan infusion 180 mg/m^2 for 90 minutes, bolus application 5-FU 400 mg/m^2 followed by 46h infusion of 5-FU 2400 mg/m^2)
  Other Names: all brands of gemcitabine and FOLFIRINOX components are allowed
Radiation: Radiotherapy, 28 x 1.8 Gy — Radiotherapy combined with chemotherapy starts on day 1 of chemotherapy. Radiation volume is restricted to macroscopic visual tumor region. Radiation is performed in 28 fractions with 1.8 Gy resulting in a total dose of 50.4 Gy.
  Arms: Induction CT, chemoradiotherapy
Drug: Chemotherapy, gemcitabine — 5 cycles of 300 mg/m^2/d gemcitabine infusions and than 3 administrations of 1000 mg/m^2/d
  Other Names: all brands of gemcitabine are allowed
  Arms: Induction CT, chemoradiotherapy
Drug: Chemotherapy with gemcitabine or FOLFIRINOX according to induction chemotherapy — Chemotherapeutic administration started with during induction chemotherapy is continued; Gemcitabine: 3 cycles a 3 administrations of 1000 mg/m^2/d gemcitabine infusions FOLFIRINOX: 6 cycles
  Other Names: all brands of gemcitabine and FOLFIRINOX components are allowed
  Arms: Induction CT, chemotherapy

SUMMARY:
This randomized trial examines the effectiveness of chemoradiotherapy compared to chemotherapy alone after induction chemotherapy with 3 cycles of gemcitabine or 6 cycles of FOLFIRINOX in patients with locally advanced, non resectable and non-metastatic pancreatic cancer. Chemotherapeutic agent in chemoradiotherapy is gemcitabine administered in 5 cycles, the agent and its administration for sole chemotherapy is determined by induction chemotherapy. Operability of tumor is evaluated at week 11 after randomisation. Patients will be followed for the duration of therapy and for 5 years after the last study treatment. Overall survival at the end of follow up is defined as primary endpoint. Secondary endpoints are tumor-free survival, rate of local recurrence or local progression, rate of distant metastasis, acute and late toxicity of the chemoradiotherapy, quality of life, rate of remission, rate of curative resections (R0) after chemotherapy and chemoradiotherapy. It is planned to include a total number of 830 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* histologically confirmed adenocarcinoma of the pancreas
* no evidence of distant metastasis based on computed tomography of the thorax and abdomen
* non resectable pancreatic cancer
* no evidence of peritoneal carcinosis
* ECOG-performance status ≤ 2
* signed study-specific consent form prior to therapy

Exclusion Criteria:

* fertile patients who refuse effective contraception during study treatment
* synchron second malignant neoplasm except basal cell carcinoma of the skin and carcinoma in situ of the cervix after curative therapy
* the Inclusion of patients with prior or concurrent malignancy (≤ 5 years prior to enrolment in study) must be discussed
* chronic inflammatory disease of the intestine
* known allergic reactions on study medication
* on-treatment participation on other trials
* insufficient liver function: Bilirubin > 2,0 mg/dl; SGOT, SGPT, alkaline phosphatase, gGT more than 3 times upper limit of normal (after Stent implantation in case of obstructive jaundice); cirrhosis of the liver Child B and C
* insufficient bone marrow function: WBC < 3,0 x 10^9/l, Platelets > 100 x 10^9/l
* serum creatinine > 1,5 mg/dl, creatinin clearance < 60ml/min (or comparable test)
* preexisting uncontrolled cardiac disease, signs of cardiac failure, or rhythm disturbances requiring therapy, myocardial infarction within the past 6 months, unstable angina pectoris, congestive heart failure, New York Heart Association (NYHA) class III or IV heart disease
* neurological and/or psychiatric diseases: stroke, dementia, epilepsy, psychosis
* active intractable or uncontrollable infection, HIV-infection
* prior radiotherapy or chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 830 (Estimated)
Dates: Start 2013-04-04 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Overall survival | Participants will be followed for the duration of therapy and for 5 years after the last study treatment

SECONDARY OUTCOMES:
Tumor-free survival | Participants will be followed for the duration of therapy and for 5 years after the last study treatment
rate of local recurrence or local progression | Participants will be followed for the duration of therapy and for 5 years after the last study treatment
Rate of distant metastasis | Participants will be followed for the duration of therapy and for 5 years after the last study treatment
Acute and late toxicity of the chemoradiotherapy | Participants will be followed for the duration of therapy and for 5 years after the last study treatment
Rate of remission | Participants will be followed for the duration of therapy and for 5 years after the last study treatment
Rate of curative resections (R0) after chemotherapy and chemoradiotherapy | Participants will be followed for the duration of therapy and for 5 years after the last study treatment
Changes in Quality of life | Participants will be followed for the duration of therapy and for 5 years after the last study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Fietkau, MD, Principal Investigator — Strahlenklinik, Universitätsklinikum Erlangen
Locations (23):
- Germany (23):
  - Bayreuth, Klinikum, Bayreuth
  - Bochum, Augusta-Kranken-Anstalt, Hämatologie/Onkologie, Bochum
  - Bochum, St. Josef-Hospital, Bochum
  - Köln Universitätsklinikum, Cologne
  - Dresden Onkologische Gemeinschaftspraxis, Dresden
  - Erlangen Universitätsklinikum, Erlangen
  - Frankfurt/Main Universitätsklinikum, Frankfurt am Main
  - Freiburg Universitätsklinikum, Freiburg im Breisgau
  - Göttingen Universitätsmedizin, Göttingen
  - Halle St. Elisabeth und St. Barbara Krankenhaus, Halle
  - Heilbronn SLK-Kliniken, Heilbronn
  - Jena Universitätsklinikum, Jena
  - Leer MVM, Leer
  - Leipzig UCCL, Leipzig
  - Magdeburg Universitätsklinikum, Magdeburg
  - Magdeburg Klinikum, Magdeburg
  - Mannheim Universitätsmedizin, Mannheim
  - München Großhadern LMU, München
  - Münster Universitätsklinikum, Münster
  - Oldenburg Pius Hospital, Oldenburg
  - Regensburg Krankenhaus Barmherzige Brüder, Regensburg
  - Regensburg Universitätsklinikum, Regensburg
  - Würzburg CCC Mainfranken, Würzburg

REFERENCES:
- [Derived] Fietkau R, Ghadimi M, Grutzmann R, Wittel UA, Jacobasch L, Uhl W, Croner RS, Bechstein WO, Neumann UP, Waldschmidt D, Boeck S, Moosmann N, Reinacher-Schick AC, Golcher H, Adler W, Semrau S, Lubgan D, Kallies A, Hecht M, Tischoff I, Tannapfel A, Frey B, Oettle H; CONKO Study Group. Benefit of Chemoradiotherapy Versus Chemotherapy After Induction Therapy for Conversion of Unresectable Into Resectable Pancreatic Cancer: The Randomized CONKO-007 Trial. J Clin Oncol. 2025 Oct 20;43(30):3266-3278. doi: 10.1200/JCO-24-01502. Epub 2025 Aug 13. PMID 40802908
- [Derived] Wittel UA, Lubgan D, Ghadimi M, Belyaev O, Uhl W, Bechstein WO, Grutzmann R, Hohenberger WM, Schmid A, Jacobasch L, Croner RS, Reinacher-Schick A, Hopt UT, Pirkl A, Oettle H, Fietkau R, Golcher H. Consensus in determining the resectability of locally progressed pancreatic ductal adenocarcinoma - results of the Conko-007 multicenter trial. BMC Cancer. 2019 Oct 22;19(1):979. doi: 10.1186/s12885-019-6148-5. PMID 31640628